CLINICAL TRIAL: NCT05474443
Title: Comparison of Instrument Assisted Soft Tissue Mobilization and Myofascial Gun in Upper Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01217 Hafsa
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Postural; Defect
Keywords: Upper Cross Syndrome; Instrument Assisted Soft Tissue Mobilization; Myofascial gun
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Intervention Model Description: 30 participants were recruited in study and divided into two groups. Group A was given intervention with Instrument Assisted Soft Tissue Mobilization and Group B with Myofascial gun
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial gun with Conventional therapy (Experimental): • Myofascial gun was applied over the Upper Trapezius muscle for 5 minutes. In the first two sessions frequency was set to 1-2 then increased to next two sessions 3-4 and so on.
  Interventions: Other: Myofascial gun with conventional therapy
- Instrument Assisted Soft Tissue Mobilization with Conventional therapy (Active Comparator): Graston's tool moved over the skin on upper trapezius muscle from its origin to insertion at 45 degree. conventional therapy applied with Thermotherapy, upper trapezius, levator scapulae and pectoralis major stretching and cryotherapy at the end
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization with Conventional therapy

INTERVENTIONS:
Other: Myofascial gun with conventional therapy — MYofascial gun was applied for the duration of 5 minutes over upper trapezius muscle. every week, on first two sessions frequency was set to 1-2 then for next two 3-4 and so on conventional therapy Hot Pack applied at the beginning of session for 10 minutes Muscle stretching of Upper Trapezius, Levator Scapulae and Pectoralis Major applied with holding time 20 seconds and 4 repetitions.
  Cold pack was applied at the end of the session for few minutes
  Arms: Myofascial gun with Conventional therapy
Other: Instrument Assisted Soft Tissue Mobilization with Conventional therapy — Graston's tool was applied over upper trapezius muscle from its origin to insertion kept at the angle of 45 Conventional Therapy Hot pack 10mins Upper Trapezius, Levator scapule and Pectoralis major muscle stretching(20s hold and 4 reps) Cold pack for few minutes
  Arms: Instrument Assisted Soft Tissue Mobilization with Conventional therapy

SUMMARY:
To compare the effects of Instrument Assisted Soft Tissue Mobilization and Myofascial gun in Upper Cross Syndrome

DETAILED DESCRIPTION:
Upper Cross Syndrome is a very common postural abnormality developed due to prolong slouched postures in desk jobs and also in students. Janda explained it that it is simultaneous presence of Forward Head Posture and protracted shoulders.

This includes weakness of lower and middle trapezius, deep neck flexors, rhomboids and serratus anterior. It also includes tightness of upper trapezius, Sternocleidomastoid, Pectoralis major and minor. The simultaneous occurrence of FHP and rounded shoulder is nothing but upper crossed syndrome.

Upper Trapezius is the primary muscle that is involved in Upper Cross Syndrome. Instrument Assisted Soft Tissue Mobilization is applied over the tight muscles to improve muscle length to its normal length. It is applied from origin to insertion with some pressure to apply compression on the muscle.

Myofascial gun is a recent technology that can be applied by the clinician and also by the affected person for self mobilization. They provide varying amount of frequencies through various shaped heads according to the area they are used,

ELIGIBILITY:
Inclusion Criteria:

• Patients with forward head posture and upper crossed syndrome

Exclusion Criteria:

* Congenital anomalies of shoulder
* Malalignment/previous fracture of clavicle
* Malignancy and Tuberculosis of spine
* Pigeon and Barrel chest

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4th week
  Changes from baseline Numeric pain Rating Scale is used to objectively assess musculoskeletal pain as marked by the patient. It is a 10 point scale from 0 to 10. 0 depicts no pain at all and 10 shows worst pain ever felt. It was measured at baseline and after 4 weeks of the intervention
Tragus to wall distance test | 4th week
  Changes from baseline Tragus to wall distance test is used to measure Forward Head Posture. The subject stands 10cm away from wall and then with the help of a ruler the distance from tragus of ear to wall is measured. If the distance was more than 9.5 cm then it was considered as forward head posture. it was measured at baseline and after 4 weeks of intervention
Neck Disability Index | 4th week
  Changes from baseline NDI is the most widely used instrument for assessing self-rated disability in patients with neck pain. The NDI is a self-report questionnaire with 10-items. The response to each item is rated on a 6-point scale from 0 (no disability) to 5 (complete disability). The numeric responses for each item are summed for a total score ranging between 0 and 50. Most of the subjects did not know how to drive so their total score was taken from 45. The questionnaire was filled by the subjects at basline and after 4 weeks of the intervention
Inclinometer | 4th week
  Changes from baseline Bubble inclinometers are portable, lightweight, inexpensive and require training. With the movement of neck the ink in the inclinometer moves and the level of ink gives the measure of the range of motion. For flexion, extension and lateral flexion of cervical Range of motion in sitting position and inclinometer was positioned at the top of head in sagittal plane. For rotations the subject was in supine position and inclinometer was placed over the forehead. Cervical ranges of motions were measured at baseline and then after 4 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No